CLINICAL TRIAL: NCT07178587
Title: Evaluating the roLe of Multiplexed PET Imaging in the Detection and Staging of hepatocellulaR Carcinoma and gAstro-entero-pancreatic Tumors: a Basket Diagnostic Performance Study
Brief Title: Evaluating the roLe of Multiplexed PET Imaging in the Detection and Staging of hepatocellulaR Carcinoma and gAstro-entero-pancreatic Tumors
Acronym: ELMIRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC24_0563
Record Dates: First submitted 2025-08-18; First posted 2025-09-17 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Hepatocellular Carcinoma (HCC); Gastro-Entero-Pancreatic Tumors (GEPs)
Keywords: Multiplexed PET; basket study; hepatocellulaR carcinoma; gAstro-entero-pancreatic tumors
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: No randomization but patients will be separated in two baskets regarding their pathologies (HCC or GEP-NET)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basket HCC (Other): Fifteen patients with HCC will be enrolled in either cohort 1 (10 patients from the University Hospital of Nantes and Beaujon Hospital) or cohort 3 (2 patients from the University Hospital of Brest for the ancillary study).
  Interventions: Diagnostic Test: Single tracer PET/CT; Diagnostic Test: Multiplexed PET-CT
- Basket GEP-NET (Other): Thirteen patients with GEP-NET will form cohort 2 (10 patients from the University Hospital of Nantes and Beaujon Hospital).
  Interventions: Diagnostic Test: Single tracer PET/CT; Diagnostic Test: Multiplexed PET-CT

INTERVENTIONS:
Diagnostic Test: Single tracer PET/CT — Single tracer PET/CT for the HCC patients : one with [18F]FDG and one with [18F]F-choline Single tracer PET/CT for the GEP-NET patients : one with [68Ga]Ga-DOTATOC and one with [18F]FDG
Diagnostic Test: Multiplexed PET-CT — Multiplexed PET-CT for HCC patients : [18F]FDG + [18F]F-choline. Multiplexed PET-CT for GEP-NET patients : [18F]FDG + [68Ga]Ga-DOTATOC. The PET scans must be performed in any order and at least 24 hours apart.

SUMMARY:
Precision medicine is a major goal in oncology. It aims to tailor treatments to the specific characteristics of each patient's tumor. This approach makes it possible to identify unique therapeutic targets and select the therapeutic alternative that specifically targets the abnormalities identified. Positron emission tomography (PET) plays a key role in this approach by providing detailed functional imaging of tumors in a non-invasive way. Usually, one radio-tracer is used to perform PET. Depending on the type of tumor, each tracer is carefully selected for its specific behavior and characteristics. However, it may be useful to perform several PET scans with different tracers, each providing different information, for the initial staging and therapeutic management of patients. Hepatocellular carcinoma (HCC), the most common form of liver cancer and the third leading cause of cancer-related death, requires precise imaging for optimal treatment selection. [18F]F-choline PET is often preferred for the initial detection of well-differentiated HCC and local recurrence, while [18F]FDG (fluorodésoxyglucose) PET is more useful for aggressive forms of HCC and for assessing metastases. Similarly, gastro-entero-pancreatic tumors (GEP-NETs), a type of neuroendocrine tumor found in the gastrointestinal tract and pancreas, also benefit from tailored imaging approaches. GEP-NETs commonly express somatostatin receptors, which are effectively targeted by [68Ga]Ga-DOTATOC PET to enhance diagnostic accuracy and staging, particularly in well-differentiated lesions. Conversely, [18F]FDG PET is valuable for imaging GEP-NETs with high metabolic activity, providing insight into tumor aggressiveness and proliferation. The combined use of [18F]FDG PET and [18F]F-choline PET in HCC, as well as [68Ga]Ga-DOTATOC PET and [18F]FDG PET in GEP-NETs, provides complementary information that helps to comprehensively characterize the tumor, guide treatment decisions, and monitor therapeutic response.

In this context, a highly innovative way using multiplexed PET imaging offers potential for targeted therapy and precision medicine. The aim of this study is to evaluate the use of simultaneous dual-tracer PET imaging with a staggered injection (referred to here as multiplexed PET), combining [18F]FDG and [18F]F-choline in HCC, and [68Ga]Ga-DOTATOC and [18F]FDG in GEP-NETs as compared to both pairs of single PET.

ELIGIBILITY:
Inclusion Criteria:

* - Men or women ≥ 18 years
* Written informed consent
* Affiliation with French social security system or beneficiary from such system
* ECOG (Eastern Cooperative Oncology Group) performance ≤ 2
* Presence of at least one morphological evaluable lesion according to RECIST 1.1 using contrast CT (computer tomography)/MRI (Magnetic Resonance Imaging) (must be performed within 6 months before inclusion)
* Willing and able to follow scheduled visits and study procedure
* Cohort 1 and 3: Child-Pugh A for cirrhotic patients (initial diagnosis, suspected relapse or progression) with histologically proven diagnosis. Albumin > 28 g/L, total bilirubin < 35 µM/L, TP>50%. The biopsy may have been performed at any point, without time limitations before inclusion.
* Cohort 2: GEP-NET (initial diagnosis, suspected relapse or progression) with histologically proven with liver metastases and/or pancreatic involvement. The biopsy may have been performed at any point, without time limitations before inclusion.
* Women must meet one of the following criteria at the time of inclusion:

  * present a negative pregnancy test (blood test) before receiving the first dose of test drug and use highly1 effective contraceptive measures for a duration of 6 months after the multiplexed PET Scan
  * or be post-menopausal (aged over 50 with amenorrhea for at least 12 months after stopping all exogenous hormone treatments);
  * or (if under 50 years of age) have been in amenorrhea for at least 12 months after stopping exogenous hormone treatments and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels corresponding to post-menopausal levels;
  * or have undergone irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy (this operation must be documented);
* Male patients will be required to use male contraception (condoms) for a duration of 3 months after the multiplexed PET Scan ;
* Women partners will be required to use an acceptable2 contraceptive measure (as they will not receive the trial drug) for a duration of 3 months after the multiplexed PET Scan ;
* Male partners will be required to use male contraception (condoms) for a duration of 6 months after the multiplexed PET Scan.

Exclusion Criteria:

* - Known hypersensitivity to gallium-68, fluor-18 to any excipient or derivative or to radiographic contrast agents.
* Any major surgery within 4 weeks before enrollment.
* Any uncontrolled significant medical, psychiatric or surgical condition or laboratory findings that, in the opinion of the investigator, might jeopardise the subject's safety or that would limit compliance with the objectives and assessments of the study.
* Other known malignancies (except for fully-resected non-melanoma skin cancer or cervical cancer in situ) unless definitively treated and proven no evidence of recurrence for 2 years.
* Women who are pregnant or breastfeeding. A serum pregnancy test will be performed at the start of the study and within 48 hours prior to multiplexed PET scan for all female subjects of childbearing potential.
* Patient under guardianship or trusteeship.
* Patient under judicial protection.
* Patient unable to understand spoken or written French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Adverse reactions collection | until 30 minutes after first injection of the first radiophamaceutical
  Safety of the staggered injection of two radiopharmaceuticals via a single route of administration will be monitored after multiplexed radiopharmaceuticals administration and until 30 minutes after the end of the image acquisition. Adverse reactions (ARs) will be collected during that period of time.
Technical Feasibility of the imaging reconstruction | within 12 months
  Technical feasibility will be qualitatively assessed for each patient by the scientific committee at the time of reconstruction of each multiplex acquisition. An image free from artifacts interfering with visual interpretation will be considered as suitable for diagnostic evaluation.
Number of positive lesions | within 12 months
  Evaluation of the diagnostic efficacy of multiplexed PET imaging for the detection and staging of both types of tumors compared to single-radiopharmaceutical PET imaging. It will be assessed by the number positive lesions using the multiplexed approach compared to lesions detected with both single-tracer PET scans. The sensitivity of the multiplex imaging over both single-tracer PET will be calculated.
Location of positive lesions | within 12 months
  Evaluation of the diagnostic efficacy of multiplexed PET imaging for the detection and staging of both types of tumors compared to single-radiopharmaceutical PET imaging. It will be assessed by the location of positive lesions using the multiplexed approach compared to lesions detected with both single-tracer PET scans. The sensitivity of the multiplex imaging over both single-tracer PET will be calculated.
quantitative information of positive lesions | within 12 months
  Evaluation of the diagnostic efficacy of multiplexed PET imaging for the detection and staging of both types of tumors compared to single-radiopharmaceutical PET imaging. It will be assessed by the quantitative information of positive lesions using the multiplexed approach compared to lesions detected with both single-tracer PET scans. The sensitivity of the multiplex imaging over both single-tracer PET will be calculated.

SECONDARY OUTCOMES:
Visual quality of multiplexed image for clinical use | within 30 days after the first PET scan
  A global assessment will be given for each multiplex imaging for the use in clinical practice. This assessment will then be summarised and presented by basket.
  The following scoring system will be used:
  * Noise quantification : 0. No noise / 1. Moderately increased noise / 2 Highly increased noise
  * Artifact detection: 0. No artifact/ 1. Presence of non-invasive artifact / 2. Presence of invasive artifact A score of 3 or more indicates poor imaging quality.
patients' satisfaction | within 30 days after the first PET scan
  Acceptability will be assessed using an ordinal scale from 1 (very uncomfortable) to 5 (very comfortable) and a one-question survey asking participants to indicate their preference between undergoing two separate single-tracer PET scans or one multiplexed PET scan
Ki computation on each of dynamic image acquisitions | within 12 months
  Exploratory analysis for patients who agreed to have dynamic whole body acquisition : Ki (capture kinetics min-1) computation on each of dynamic image acquisitions
Tumor normalized uptake values (SUV) (Exploratory analysis) | within 12 months
  Exploratory analysis for patients who agreed to have dynamic whole body acquisition : Tumor normalized uptake values (SUV) will be determined on each imaging PET to evaluate whether dynamic PET/CT (computing tomography) imaging (including multiplexed imaging) improves lesion detection compared with static PET/CT
Vd computation on each of dynamic image acquisitions | within 12 months
  Exploratory analysis for patients who agreed to have dynamic whole body acquisition : Vd (volume of distribution) computation on each of dynamic image acquisitions

CONTACTS AND LOCATIONS:
Overall Officials: Thomas CARLIER, PhD, Study Chair — Nantes University Hospital; Yann TOUCHEFEU, MD, Study Director — Nantes University Hospital
Locations (3):
- France (3):
  - CHU Brest, Brest
  - Hopital Foch (AP-HP), Clichy
  - Chu Nantes, Nantes

IPD SHARING:
Plan to Share IPD: No